CLINICAL TRIAL: NCT02132949
Title: A Multicenter, Multinational, Phase II Study to Evaluate Perjeta in Combination With Herceptin and Standard Neoadjuvant Anthracycline-Based Chemotherapy in Patients With HER2-Positive, Locally Advanced, Inflammatory, or Early-Stage Breast Cancer
Brief Title: A Study Evaluating Pertuzumab (Perjeta) Combined With Trastuzumab (Herceptin) and Standard Anthracycline-based Chemotherapy in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Locally Advanced, Inflammatory, or Early-stage Breast Cancer
Acronym: BERENICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29217; 2014-000156-28 (EudraCT Number)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Paclitaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab (Experimental): Participants received neoadjuvant treatment with dose-dense doxorubicin and cyclophosphamide (ddAC), with administration of doxorubicin 60 milligrams per square meter (mg/m^2) intravenously (IV) once every 2 weeks (q2w) and cyclophosphamide 600mg/m^2 IV q2w for 4 cycles, followed by paclitaxel 80mg/m^2 IV once weekly (qw) for 12 weeks. Pertuzumab (840 milligrams [mg] IV loading dose then 420mg IV q3w) and trastuzumab (8 milligrams per kilogram [mg/kg] IV loading dose then 4mg/kg IV q3w) were administered along with paclitaxel for 4 cycles (8 cycles of chemotherapy in total prior to surgery). Following surgery, participants received adjuvant treatment with pertuzumab and trastuzumab IV q3w (up to 13 cycles), for a total of 17 cycles of pertuzumab and trastuzumab therapy during the study. Radiotherapy and adjuvant hormonal therapy were also given as clinically indicated. Following treatment completion/discontinuation, participants were followed for safety and efficacy for up to 5 years.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab (Experimental): Participants received neoadjuvant treatment with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC), with administration of 5-fluorouracil 500mg/m^2 intravenously (IV) q3w, epirubicin 100mg/m^2 IV q3w, and cyclophosphamide 600mg/m^2 IV q3w for 4 cycles, followed by docetaxel (with starting dose of 75mg/m^2 in Cycle 5, then 100mg/m^2 for Cycles 6-8) q3w for 4 cycles. Pertuzumab (840 mg IV loading dose then 420mg IV q3w) and trastuzumab (8 mg/kg IV loading dose then 4mg/kg IV q3w) were given along with doectaxel for 4 cycles (8 cycles of chemotherapy in total prior to surgery). Following surgery, participants received adjuvant treatment with pertuzumab and trastuzumab IV q3w (up to 13 cycles), for a total of 17 cycles of pertuzumab and trastuzumab therapy during the study. Radiotherapy and adjuvant hormonal therapy were also given as clinically indicated. Following treatment completion/discontinuation, participants were followed for safety and efficacy for up to 5 years.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Epirubicin; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive 5-fluorouracil 500 mg/m^2 IV on Day 1 of each cycle q3w.
  Arms: Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Drug: Cyclophosphamide — Participants will receive cyclophosphamide 600 milligrams per square meter (mg/m^2) intravenous (IV) given on Day 1 of each cycle q2w.
Drug: Docetaxel — Participants will receive docetaxel at a starting dose of 75 mg/m^2 IV for the first cycle and the dose may be escalated to 100 mg/m^2 for subsequent cycles q3w.
  Arms: Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Drug: Doxorubicin — Participants will receive doxorubicin 60 mg/m^2 IV on Day 1 of each cycle q2w.
  Arms: Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab
Drug: Epirubicin — Participants will receive epirubicin 100 mg/m^2 IV on Day 1 of each cycle q3w.
  Arms: Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Drug: Paclitaxel — Participants will receive paclitaxel 80 mg/m^2 IV given weekly.
  Arms: Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab
Drug: Pertuzumab — Participants will receive pertuzumab at a loading dose of 840 milligrams (mg) IV loading dose, then 420 mg IV q3w.
  Other Names: Perjeta
Drug: Trastuzumab — Participants will receive trastuzumab at a loading dose of 8 milligrams per kilogram (mg/kg) IV, then 6 mg/kg IV q3w.
  Other Names: Herceptin

SUMMARY:
This multicenter, non-randomized, open-label, phase 2 study is designed to evaluate the safety and efficacy of pertuzumab (Perjeta) in combination with trastuzumab (Herceptin) and anthracycline-based chemotherapy as neoadjuvant treatment in participants with HER2-positive locally advanced, inflammatory, or early-stage breast cancer. Each investigator will choose a treatment regimen (A or B) for all of their participants to follow. Treatment regimen A (for Cohort A) will include dose-dense doxorubicin and cyclophosphamide (ddAC), followed by paclitaxel, with pertuzumab and trastuzumab given from the start of paclitaxel. Treatment regimen B (for Cohort B) will include 5-fluorouracil, epirubicin, and cyclophosphamide (FEC), followed by docetaxel, with pertuzumab and trastuzumab given from the start of docetaxel. Participants in both cohorts will subsequently undergo surgical treatment and then resume pertuzumab and trastuzumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with locally advanced, inflammatory, or early-stage, unilateral, and histologically confirmed invasive breast cancer. Participants with inflammatory breast cancer must be able to have a core needle biopsy
* Primary tumor greater than (>) 2 centimeters (cm) in diameter, or > 5 millimeters (mm) in diameter and node-positive
* HER2-positive breast cancer confirmed by a central laboratory
* Availability of tumor tissue specimen
* Baseline LVEF greater than or equal to (>/=) 55%
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (</=) 1
* At least 4 weeks since major unrelated surgery, with full recovery
* Women of childbearing potential and male participants with partners of childbearing potential must agree to use a "highly effective" non-hormonal form of contraception or two "effective" forms of non-hormonal contraception by the patient and/or partner. Contraception must continue for the duration of study treatment and for at least 7 months after the last dose of study treatment

Exclusion Criteria:

* Metastatic disease (Stage IV) or bilateral breast cancer
* Participants who have had an incisional biopsy of the primary tumor or the primary tumor excised
* Prior breast or non-breast malignancy within 5 years prior to study entry, except for carcinoma in situ and basal cell and squamous cell carcinoma of the skin. Participants with malignancies occurring more than 5 years prior to study entry are permitted if curatively treated
* Any previous systemic therapy (including chemotherapy, immunotherapy, HER2 targeted agents, and antitumor vaccines) for cancer, or radiation therapy for cancer
* Participants with a past history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) are not allowed to enter the study if they have received any systemic therapy for its treatment or radiation therapy to the ipsilateral breast (they are allowed to enter the study if treated with surgery alone)
* High-risk participants who have received chemopreventive drugs in the past are not allowed to enter the study
* Inadequate bone marrow, renal, or liver function
* History or evidence of cardiovascular condition
* Dyspnea at rest or other diseases that require continuous oxygen therapy
* Severe, uncontrolled systemic disease
* Participants with poorly controlled diabetes or with evidence of clinically significant diabetic vascular complications
* Pregnancy or breast-feeding women
* Participants who received any investigational treatment within 4 weeks of study start
* Participants with known infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* Current chronic daily treatment with corticosteroids (dose >10 mg methylprednisolone or equivalent [excluding inhaled steroids])
* Known hypersensitivity to any of the study drugs or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- United States (24):
  - University of South Alabama; Mitchell Cancer Institute, Mobile, Alabama
  - Marin Specialty Care, Greenbrae, California
  - California Pacific Medical Center, San Francisco, California
  - MedStar Georgetown University Hospital (Lombardi Comprehensive Cancer Center), Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center., Washington D.C., District of Columbia
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Saint Lukes Hospital Cancer Institute, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Regional Cancer Care Associates LLC - Morristown, Morristown, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - MSKCC @ Commack, Commack, New York
  - MSKCC @ West Harrison, Harrison, New York
  - Mount Sinai Beth Israel Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSKC @ Rockville, Rockville Centre, New York
  - Mercy Clinic Oklahoma Communties, Inc, Oklahoma City, Oklahoma
  - Harrington Cancer Center, Amarillo, Texas
  - University of Utah; Huntsman Cancer Hospital, Salt Lake City, Utah
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - PeaceHealth St. Joseph Cancer Center, Bellingham, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Canada (6):
  - Horizon Health Network, Moncton, New Brunswick
  - Royal Victoria Hospital, Barrie, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - St Mary's Hospital Center, Montreal, Quebec
  - Hopital Sacre-Coeur Research Centre, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Denmark (3):
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Rigshospitalet; Onkologisk Klinik, København Ø
  - Vejle Sygehus; Onkologisk Afdeling, Vejle
- France (9):
  - Clinique Victor Hugo; Chimiotherapie, Le Mans
  - Centre Oscar Lambret; Cancerologie Gynecologique, Lille
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Institut Curie; Oncologie Medicale, Paris
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (5):
  - Universitätsklinikum "Carl Gustav Carus"; Frauenheilkunde und Geburtshilfe, Dresden
  - Dres.Andreas Ammon und Dirk Meyer, Göttingen
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - Klinikum rechts der Isar der TU München; Klinik und Poliklinik für Frauenheilkunde, München
  - Ruppiner Kliniken, Klinik fuer Gynaekologie und Geburtshilfe, Neuruppin
- Italy (6):
  - Asl Le-Ospedale "Vito Fazzi";U.O. Oncologia, Lecce, Apulia
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Casa Di Cura Di Alta Specialita La Maddalena; Dept. Oncologico Di Iii Livello, Palermo, Sicily
  - Ospedale Santa Maria Annunziata; Oncologia, Bagno a Ripoli, Tuscany
  - Ospedale Della Misericordia; U.O. Di Medicina Ia - Oncologia Medica, Grosseto, Tuscany
- Mexico (2):
  - Iem-Fucam, D.F.
  - Centro de Diagnóstico y Tratamiento Integral de Mama, Hospital San José Tec de Monterrey, Monterrey
- Norway (2):
  - Haukeland Universitetssjukehus; Klinisk forskningspost, Bergen
  - Oslo universitetssykehus HF, Ullevål, Kreftsenteret, Oslo
- Poland (4):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Wielkopolskie Centrum Onkologii; im. Marii Skłodowskiej-Curie, Poznan
- Portugal (4):
  - Centro Clinico Champalimaud; Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Centro Oncológico Gallego José Antonio Quiroga y Piñeiro, Servicio de Oncologia, A Coruña
  - Hospital Universitario de la Princesa; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
- United Kingdom (8):
  - Royal United Hospital; Oncology Department, Bath
  - Royal Bournemouth Hospital; Oncology, Bournemouth
  - Guys & St Thomas Hospital; Department of Oncology, London
  - Royal Marsden Hospital - Fulham; Oncology Department, London
  - Freeman Hospital; Northern Centre For Cancer Care, New Castle Upon Tyne
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Peterborough City Hospital, Edith Cavell Campus; Oncology Department, Peterborough
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Swain SM, Ewer MS, Viale G, Delaloge S, Ferrero JM, Verrill M, Colomer R, Vieira C, Werner TL, Douthwaite H, Bradley D, Waldron-Lynch M, Kiermaier A, Eng-Wong J, Dang C; BERENICE Study Group. Pertuzumab, trastuzumab, and standard anthracycline- and taxane-based chemotherapy for the neoadjuvant treatment of patients with HER2-positive localized breast cancer (BERENICE): a phase II, open-label, multicenter, multinational cardiac safety study. Ann Oncol. 2018 Mar 1;29(3):646-653. doi: 10.1093/annonc/mdx773. PMID 29253081

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 401 participants were enrolled, 199 in Cohort A and 202 in Cohort B. One participant in Cohort B who was human epidermal growth factor receptor 2 (HER2) negative and was enrolled by error, was excluded. Hence, 199 participants were included in Cohort A and 201 participants in Cohort B.
Period: Overall Study
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Started (ITT Population) | 199 | 201 (1 participant enrolled in Cohort B received Cohort A treatment (and was counted as part of Cohort B for efficacy).)
Received Any Cohort A Study Treatment (Safety Population for Cohort A) | 198 (1 participant withdrew prior to receiving any study drug.) | 1 (1 participant enrolled in Cohort B received Cohort A treatment (and was counted as part of Cohort A for safety).)
Received Any Cohort B Study Treatment (Safety Population for Cohort B) | 0 | 198 (2 participants withdrew prior to receiving any study drug.)
Underwent Surgery | 187 | 194
Completed Neoadjuvant Treatment (25 Weeks) | 182 | 189
Started Adjuvant Treatment | 181 | 190 (1 participant did not complete neoadjuvant treatment but started adjuvant treatment.)
Completed Adjuvant Treatment (Up to 39 Weeks) | 163 | 176
Started Treatment-Free Follow-Up (Up to 5 Years) (Includes participants who completed or discontinued neoadjuvant/adjuvant treatment.) | 195 | 195
Completed | 158 | 173
Not Completed | 41 | 28
Not completed — Death | 7 | 13
Not completed — Lost to Follow-up | 14 | 4
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Noncompliance | 5 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Disease Progression | 3 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Withdrew Prior to Treatment | 1 | 2
Not completed — Reason Unspecified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who were enrolled regardless of whether they received any study treatment. One participant in Cohort B who was HER2 negative and was enrolled by error was excluded from the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab | Total
Number analyzed (Participants) | 199 | 201 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.7) | 49.5 (11.5) | 49.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 200 | 399
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 46 | 70
  Not Hispanic or Latino | 147 | 114 | 261
  Unknown or Not Reported | 28 | 41 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 6
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 0 | 11
  White | 162 | 163 | 325
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 34 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Event of New York Heart Association (NYHA) Class III or IV Heart Failure During the Neoadjuvant Treatment Period
Description: Symptomatic left ventricular systolic dysfunction (otherwise referred to as heart failure) is a serious adverse event. The NYHA Functional Classification System for Heart Failure considers the patient's symptoms: Class III: Marked limitation of physical activity; Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry on any physical activity without discomfort; Symptoms of heart failure at rest; If any physical activity is undertaken, discomfort increases. The 95% CIs were calculated with the Clopper-Pearson method. Results included events with onset from first dose of pertuzumab/trastuzumab prior to surgery through the day before the first dose of any study drug after surgery. If participant withdrew without entering adjuvant period, results included all events with onset from first dose of pertuzumab/trastuzumab through 42 days after last dose of any study drug or on the day of target surgery whichever was later.
Time Frame: From day of first dose of pertuzumab or trastuzumab until the end of the neoadjuvant treatment period (as defined in the description; up to 25 weeks)
Population: Safety analysis population of all participants who received any study treatment during the neoadjuvant treatment period, grouped according to treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
percentage of participants | 1.5 [0.31 to 4.34] | 0 [0.00 to 1.85]

2. Primary Outcome: Percentage of Participants With at Least One Left Ventricular Ejection Fraction (LVEF) Significant Decline, Defined as a Drop in LVEF of at Least 10 Percentage Points From Baseline and to Below 50%, During the Neoadjuvant Treatment Period
Description: LVEF significant decline was defined as the decline in LVEF of >/= 10%-points from baseline to an LVEF of < 50%. A Confirmed LVEF Significant Decline was defined as at least two consecutive readings of significant declines in LVEF. A Single LVEF Significant Decline was defined as only one reading of a significant decline (no consecutive readings) in LVEF. The category of 'At Least one LVEF Significant Decline Event' was defined as the total of confirmed and single LVEF significant declines. The 95% confidence intervals (CIs) were calculated using the Clopper-Pearson method. Results include events with onset from the first dose of pertuzumab or trastuzumab prior to surgery through the day before the first dose of any study drug after surgery. If participant withdrew without entering adjuvant period, results included all events with onset from first dose of pertuzumab or trastuzumab through 42 days after last dose of any study drug or on the day of target surgery whichever is later.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
percentage of participants
  At Least One LVEF Significant Decline Event (Confirmed+Single) | 6.5 [3.5 to 10.9] | 2.0 [0.6 to 5.1]
  At Least One Confirmed LVEF Significant Decline | 1.0 [0.1 to 3.6] | 0.5 [0.0 to 2.8]
  At Least One Single LVEF Significant Decline | 5.5 [2.8 to 9.7] | 1.5 [0.3 to 4.4]

3. Secondary Outcome: Percentage of Participants With at Least One Event of New York Heart Association (NYHA) Class III or IV Heart Failure During the Adjuvant Treatment Period
Description: Symptomatic left ventricular systolic dysfunction (otherwise referred to as heart failure) is a serious adverse event. The NYHA Functional Classification System for Heart Failure considers the patient's symptoms: Class III: Marked limitation of physical activity; Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry on any physical activity without discomfort; Symptoms of heart failure at rest; If any physical activity is undertaken, discomfort increases. The 95% CIs were calculated with the Clopper-Pearson method. Results included events with onset from the first dose of any study drug after surgery through 42 days after the last dose of any study drug.
Time Frame: From the first dose of any study drug after surgery through 42 days after the last dose of any study drug (during the adjuvant treatment period; up to approximately 39 weeks)
Population: Safety analysis population of all participants who started and received any study treatment during the adjuvant treatment period, grouped according to treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 181 | 190
Percentage of participants | 0 [0.00 to 2.02] | 0.5 [0.01 to 2.90]

4. Secondary Outcome: Percentage of Participants With at Least One Left Ventricular Ejection Fraction (LVEF) Significant Decline, Defined as a Drop in LVEF of at Least 10 Percentage Points From Baseline and to Below 50%, During the Adjuvant Treatment Period
Description: LVEF significant decline was defined as the decline in LVEF of >/= 10%-points from baseline to an LVEF of < 50%. A Confirmed LVEF Significant Decline was defined as at least two consecutive readings of significant declines in LVEF. A Single LVEF Significant Decline was defined as only one reading of a significant decline (no consecutive readings) in LVEF. The category of 'At Least one LVEF Significant Decline Event' was defined as the total of confirmed and single LVEF significant declines. The 95% confidence intervals were calculated using the Clopper-Pearson method. Results included events with onset from the first dose of any study drug after surgery through 42 days after the last dose of any study drug.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 181 | 190
percentage of participants
  At Least One LVEF Significant Decline Event (Confirmed+Single) | 7.7 [4.3 to 12.6] | 10.5 [6.5 to 15.8]
  At Least One Confirmed LVEF Significant Decline | 2.8 [0.9 to 6.3] | 3.2 [1.2 to 6.7]
  At Least One Single LVEF Significant Decline | 5.0 [2.3 to 9.2] | 7.4 [4.1 to 12.1]

5. Secondary Outcome: Percentage of Participants With at Least One Event of New York Heart Association (NYHA) Class III or IV Heart Failure During the Treatment-Free Follow-Up Period
Description: Symptomatic left ventricular systolic dysfunction (otherwise referred to as heart failure) is a serious adverse event. The NYHA Functional Classification System for Heart Failure considers the patient's symptoms: Class III: Marked limitation of physical activity; Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV: Unable to carry on any physical activity without discomfort; Symptoms of heart failure at rest; If any physical activity is undertaken, discomfort increases. The 95% CIs were calculated with the Clopper-Pearson method.
Time Frame: From 42 days after the last dose of study treatment until the end of treatment-free follow-up (up to 5 years)
Population: Safety analysis population of all participants who received any study treatment during the study, grouped according to treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
Percentage of participants | 0 [0.00 to 1.84] | 0.5 [0.01 to 2.78]

6. Secondary Outcome: Percentage of Participants With at Least One Left Ventricular Ejection Fraction (LVEF) Significant Decline, Defined as a Drop in LVEF of at Least 10 Percentage Points From Baseline and to Below 50%, During the Treatment-Free Follow-Up Period
Description: LVEF significant decline was defined as the decline in LVEF of >/= 10%-points from baseline to an LVEF of < 50%. A Confirmed LVEF Significant Decline was defined as at least two consecutive readings of significant declines in LVEF. A Single LVEF Significant Decline was defined as only one reading of a significant decline (no consecutive readings) in LVEF. The category of 'At Least one LVEF Significant Decline Event' was defined as the total of confirmed and single LVEF significant declines. The 95% confidence intervals were calculated using the Clopper-Pearson method.
Time Frame: From 42 days after the last dose of study treatment until the end of treatment-free follow-up (up to 5 years)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
Percentage of participants
  At Least One LVEF Significant Decline Event (Confirmed+Single) | 6.0 [3.2 to 10.3] | 3.5 [1.4 to 7.1]
  At Least One Confirmed LVEF Significant Decline | 3.0 [1.1 to 6.4] | 1.0 [0.1 to 3.6]
  At Least One Single LVEF Significant Decline | 3.0 [1.1 to 6.4] | 2.5 [0.8 to 5.8]

7. Secondary Outcome: Overview of the Number of Participants With at Least One Adverse Event During the Neoadjuvant Period
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. The terms "severe" and "serious" are not synonymous with respect to an AE. Severity refers to the intensity of an AE (rated according to NCI-CTCAE v4.0 criteria or, if not listed, the following scale: Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to AE), whereas a serious AE (SAE) is a significant medical event (per standard criteria). Severity and seriousness needed to be independently assessed for each AE that was recorded. Selected AEs for reporting included heart failure (NYHA Class II/III/IV) and asymptomatic declines in LVEF (reported as an AE with the term of ejection fraction decreased). In the results table, multiple occurrences of the same AE in one individual were counted only once. Any AE includes all serious and non-serious AEs.
Time Frame: From first dose of any study drug prior to surgery through the day before the first dose of study drug after surgery (up to 25 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
Participants
  Any Adverse Event (AE) | 198 | 198
  NCI-CTCAE Grade 3-5 AE | 99 | 108
  Serious AE | 45 | 52
  Deaths | 0 | 0
  Ejection Fraction Decreased (Any Grade) | 14 | 7
  Heart Failure (Any Grade) | 4 | 0

8. Secondary Outcome: Overview of the Number of Participants With at Least One Adverse Event During the Adjuvant Period
Description: as for outcome 7
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 181 | 190
Participants
  Any Adverse Event (AE) | 171 | 171
  NCI-CTCAE Grade 3-5 AE | 23 | 40
  Serious AE | 15 | 17
  Deaths | 0 | 0
  Ejection Fraction Decreased (Any Grade) | 15 | 20
  Heart Failure (Any Grade) | 0 | 2

9. Secondary Outcome: Overview of the Number of Participants With at Least One Adverse Event During the Treatment-Free Follow-Up Period
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (rated according to NCI-CTCAE v4.0 criteria or, if not listed, the following scale: Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to AE), and a serious AE (SAE) is a significant medical event (per standard criteria). Severity and seriousness were independently assessed for each AE. Selected AEs for reporting included heart failure (NYHA Class II/III/IV) and asymptomatic declines in LVEF (reported as ejection fraction decreased). During TFFU, only heart failure, pregnancies, and non-breast-related second primary malignancies, irrespective of causal relationship with study treatment, and drug-related SAEs were reported. Multiple occurrences of the same AE in 1 subject were counted only once.
Time Frame: From 42 days after the last dose of study treatment until the end of treatment-free follow-up (TFFU; up to 5 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 198
Participants
  Any Adverse Event (AE) | 3 | 7
  NCI-CTCAE Grade 3-5 AE | 2 | 5
  Serious AE | 3 | 7
  Deaths | 7 | 13
  Ejection Fraction Decreased (Any Grade) | 1 | 1
  Heart Failure (Any Grade) | 0 | 1

10. Secondary Outcome: Percentage of Participants Positive for Anti-Therapeutic Antibodies (ATAs) to Pertuzumab at Baseline and Anytime Post-Baseline
Description: ATAs to pertuzumab in serum samples were detected using a validated bridging enzyme-linked immunosorbent assay (ELISA) method. This analysis only included participants with an ATA assay result from a baseline sample and/or at least one post-baseline sample.
Time Frame: Screening (baseline) then prior to pertuzumab infusion (Hour 0) in Cycles 5, 14, 18 thereafter anytime between Cycle 8 Day 21 and surgery, up to treatment completion visit (cycle length=2-3 weeks; up to approximately 1 year, 3 months)
Population: This analysis only included participants with an ATA assay result from a baseline sample and/or at least one post-baseline sample.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 201
Percentage of participants
  At Baseline: number analyzed (Participants) | 190 | 191
  At Baseline | 1.6 | 2.1
  Anytime Post-Baseline: number analyzed (Participants) | 195 | 197
  Anytime Post-Baseline | 4.6 | 3.6

11. Secondary Outcome: Percentage of Participants With Total Pathologic Complete Response (tpCR), Evaluated After Surgery
Description: Total pathologic complete response (tpCR) was the pCR based on tumor and nodal staging (i.e., histological confirmation of pCR in breast and nodes at surgery) and was defined as the absence of any residual invasive cancer in the breast and the absence of any metastatic cells in the regional lymph nodes (i.e., ypT0/is ypN0 tpCR). Participants who did not undergo surgery or did not have a valid pCR assessment were considered non-responders in the analysis. The 95% CIs were calculated using the Clopper-Pearson method.
Time Frame: After completion of neoadjuvant treatment and surgery (up to 25 weeks)
Population: ITT population: included all participants who were enrolled regardless of whether they received any study treatment, grouped according to the arm to which a participant was enrolled.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 201
Percentage of participants | 61.8 [54.67 to 68.59] | 60.7 [53.58 to 67.49]

12. Secondary Outcome: Percentage of Participants With Clinical Response as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 During the Neoadjuvant Treatment Period
Description: The clinical response rate was defined as the percentage of participants in the ITT population who achieved a complete response (CR) or partial response (PR) prior to surgery, according to RECIST v1.1. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the longest diameter compared to Baseline. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient (20%) increase to qualify for disease progression, in addition to no new target lesions. Progressive Disease (PD): at least a 20% increase in the sum of the longest diameter, taking as reference the smallest sum of the longest diameter observed at previous tumor assessment, or the appearance of any new lesions. Participants were classified as missing or unevaluable if no assessments were measured prior to surgery on the ipsilateral breast. The 95% CIs were calculated using the Clopper-Pearson method; they were only calculated for responses (not for missing or unevaluable data).
Time Frame: From Baseline until disease progression or death due to any cause up to 24 weeks (during the neoadjuvant treatment period; assessed on Day 1 of Cycles 1-8 [cycle length=2-3 weeks])
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 201
Percentage of participants
  Clinical Response Rate (CR+PR) | 67.3 [60.35 to 73.80] | 60.2 [53.07 to 67.02]
  Complete Response (CR) | 39.7 [32.85 to 46.86] | 23.9 [18.16 to 30.39]
  Partial Response (PR) | 27.6 [21.55 to 34.41] | 36.3 [29.67 to 43.38]
  Stable Disease (SD) | 7.0 [3.90 to 11.52] | 10.0 [6.18 to 14.95]
  Progressive Disease (PD) | 0.5 [0.01 to 2.77] | 1.0 [0.12 to 3.55]
  Missing or Unevaluable | 25.1 [NA to NA] — 95% CIs were only calculated for responses, not for missing or unevaluable data. | 28.9 [NA to NA] — 95% CIs were only calculated for responses, not for missing or unevaluable data.

13. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Event-Free Survival (EFS) at 1 to 5 Years, Determined by the Investigator According to RECIST v1.1
Description: The Kaplan-Meier method was used to estimate the percentage of participants who were event-free at landmark timepoints. Event-free survival (EFS) was defined as the time from enrollment to the first occurrence of progressive disease (PD), relapse, or death from any cause, with tumor evaluations performed by the investigator according to RECIST v1.1. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) were not counted as progressive disease or relapse. Participants who withdrew from the study without documented progression or relapse and for whom there existed evidence that evaluations had been made, were censored at the date of the last assessment at which the participant was known to be free from progressive disease or relapse. Participants with no tumor evaluations after baseline were censored at the date of enrollment plus 1 day.
Time Frame: At 1, 2, 3, 4, and 5 years
Population: ITT population: included all participants who were enrolled regardless of whether they received any study treatment, grouped according to the arm to which a participant was enrolled. The number analyzed per timepoint represents the number of participants remaining at risk at that timepoint.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 201
Estimate of percentage of participants
  1 Year: number analyzed (Participants) | 191 | 190
  1 Year | 98.47 [96.75 to 100.00] | 97.48 [95.29 to 99.66]
  2 Years: number analyzed (Participants) | 176 | 180
  2 Years | 95.80 [92.94 to 98.65] | 92.86 [89.25 to 96.46]
  3 Years: number analyzed (Participants) | 163 | 174
  3 Years | 93.58 [90.06 to 97.10] | 90.78 [86.72 to 94.84]
  4 Years: number analyzed (Participants) | 154 | 172
  4 Years | 92.39 [88.55 to 96.23] | 89.73 [85.47 to 94.00]
  5 Years: number analyzed (Participants) | 96 | 141
  5 Years | 90.84 [86.48 to 95.20] | 89.20 [84.84 to 93.57]

14. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Invasive Disease-Free Survival (iDFS) at 1 to 4 Years, Determined by the Investigator According to RECIST v1.1
Description: The Kaplan-Meier method was used to estimate the percentage of participants who were event-free at landmark timepoints. Invasive disease-free survival (iDFS) was defined as the time from the first date of no disease (the date of surgery) to the first documentation of progressive invasive disease, relapse, or death, with tumor evaluations performed by the investigator according to RECIST v1.1. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) were not counted as progressive disease or relapse. Participants who withdrew from the study without documented progression or relapse and for whom there existed evidence that evaluations had been made, were censored at the date of the last assessment at which the participant was known to be alive and disease-free. Participants with no postbaseline information and participants who did not undergo surgery were excluded from the analysis.
Time Frame: At 1, 2, 3, and 4 years
Population: ITT population: included all participants who were enrolled regardless of whether they received any study treatment, grouped according to the arm to which a participant was enrolled. Participants with no post-baseline information and those who did not undergo surgery were excluded from the analysis. The number analyzed per timepoint represents the number of participants remaining at risk at that timepoint.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 187 | 194
Estimate of percentage of participants
  1 Year: number analyzed (Participants) | 180 | 184
  1 Year | 98.91 [97.41 to 100.00] | 96.34 [93.68 to 99.00]
  2 Years: number analyzed (Participants) | 167 | 178
  2 Years | 95.57 [92.57 to 98.57] | 94.25 [90.94 to 97.55]
  3 Years: number analyzed (Participants) | 158 | 171
  3 Years | 94.42 [91.06 to 97.78] | 91.06 [87.00 to 95.11]
  4 Years: number analyzed (Participants) | 131 | 168
  4 Years | 92.60 [88.72 to 96.48] | 91.06 [87.00 to 95.11]

15. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Overall Survival (OS) at 1 to 5 Years
Description: The Kaplan-Meier method was used to estimate the percentage of participants who were event-free at landmark timepoints. Overall survival (OS) was defined as the time from enrollment to death from any cause. Participants who were alive or lost to follow-up were censored at their last known date in the study. Participants with no post-baseline assessments were censored at the date of enrollment plus 1 day.
Time Frame: At 1, 2, 3, 4, and 5 years
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
Number analyzed (Participants) | 199 | 201
Estimate of percentage of participants
  1 Year: number analyzed (Participants) | 193 | 194
  1 Year | 99.48 [98.48 to 100.00] | 100.00 [100.00 to 100.00]
  2 Years: number analyzed (Participants) | 183 | 190
  2 Years | 98.96 [97.52 to 100.00] | 97.94 [95.94 to 99.94]
  3 Years: number analyzed (Participants) | 176 | 185
  3 Years | 97.86 [95.78 to 99.94] | 96.38 [93.74 to 99.01]
  4 Years: number analyzed (Participants) | 171 | 180
  4 Years | 97.86 [95.78 to 99.94] | 94.81 [91.68 to 97.94]
  5 Years: number analyzed (Participants) | 158 | 177
  5 Years | 96.10 [93.26 to 98.94] | 93.75 [90.33 to 97.17]

ADVERSE EVENTS:
Time Frame: From first dose of any study drug until the end of treatment-free follow-up (up to 6 years, 1 month)
Arm/Group | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab
All-Cause Mortality (participants affected / at risk) | 7/199 | 13/198
Serious Adverse Events (participants affected / at risk) | 56/199 | 66/198
Other Adverse Events (participants affected / at risk) | 197/199 | 198/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab (N=199) | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab (N=198)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 11 (11) | 27 (28)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 4 (4)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 11 (12)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 4 (5)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
BREAST CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 3 (3) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
MASTITIS (Infections and infestations) | 2 (4) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 7 (7)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 2 (2) | 3 (3)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
WOUND DECOMPOSITION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 5 (5) | 5 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (3) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBELLAR SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 0 (0)
BREAST HAEMATOMA (Reproductive system and breast disorders) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ddAC, Paclitaxel, Pertuzumab, Trastuzumab (N=199) | Cohort B: FEC, Docetaxel, Pertuzumab, Trastuzumab (N=198)
ANAEMIA (Blood and lymphatic system disorders) | 56 (65) | 64 (78)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 10 (10)
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 (5) | 11 (16)
NEUTROPENIA (Blood and lymphatic system disorders) | 43 (54) | 31 (43)
PALPITATIONS (Cardiac disorders) | 10 (12) | 11 (12)
VERTIGO (Ear and labyrinth disorders) | 4 (4) | 10 (11)
DRY EYE (Eye disorders) | 13 (13) | 13 (13)
LACRIMATION INCREASED (Eye disorders) | 20 (20) | 37 (37)
VISION BLURRED (Eye disorders) | 13 (16) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (12) | 27 (38)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 (17) | 31 (33)
CONSTIPATION (Gastrointestinal disorders) | 73 (87) | 78 (90)
DIARRHOEA (Gastrointestinal disorders) | 143 (207) | 141 (238)
DRY MOUTH (Gastrointestinal disorders) | 13 (13) | 17 (18)
DYSPEPSIA (Gastrointestinal disorders) | 40 (46) | 35 (42)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 27 (27) | 6 (6)
HAEMORRHOIDS (Gastrointestinal disorders) | 19 (20) | 22 (26)
MOUTH ULCERATION (Gastrointestinal disorders) | 5 (5) | 15 (16)
NAUSEA (Gastrointestinal disorders) | 144 (181) | 142 (196)
ODYNOPHAGIA (Gastrointestinal disorders) | 7 (7) | 10 (13)
STOMATITIS (Gastrointestinal disorders) | 49 (53) | 56 (73)
VOMITING (Gastrointestinal disorders) | 46 (57) | 71 (107)
ASTHENIA (General disorders) | 41 (72) | 85 (130)
CHILLS (General disorders) | 12 (14) | 4 (4)
FATIGUE (General disorders) | 125 (151) | 81 (119)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (8) | 21 (24)
MUCOSAL INFLAMMATION (General disorders) | 46 (55) | 77 (106)
OEDEMA (General disorders) | 5 (5) | 10 (10)
OEDEMA PERIPHERAL (General disorders) | 22 (25) | 28 (35)
PAIN (General disorders) | 16 (18) | 6 (6)
PYREXIA (General disorders) | 39 (45) | 39 (53)
CONJUNCTIVITIS (Infections and infestations) | 10 (10) | 16 (18)
INFLUENZA (Infections and infestations) | 8 (9) | 14 (16)
NASOPHARYNGITIS (Infections and infestations) | 21 (30) | 33 (40)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 10 (10)
PHARYNGITIS (Infections and infestations) | 8 (8) | 13 (14)
RHINITIS (Infections and infestations) | 7 (8) | 18 (19)
SINUSITIS (Infections and infestations) | 11 (12) | 9 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 25 (28) | 6 (7)
URINARY TRACT INFECTION (Infections and infestations) | 32 (36) | 10 (11)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 38 (42) | 35 (50)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 17 (18) | 12 (14)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 36 (36) | 58 (59)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 15 (19) | 13 (15)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 14 (18) | 11 (12)
EJECTION FRACTION DECREASED (Investigations) | 22 (27) | 22 (27)
LYMPHOCYTE COUNT DECREASED (Investigations) | 12 (15) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 18 (22) | 19 (26)
WEIGHT DECREASED (Investigations) | 19 (19) | 13 (13)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 22 (29) | 6 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 40 (42) | 49 (59)
DEHYDRATION (Metabolism and nutrition disorders) | 10 (14) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 16 (18) | 6 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 73 (96) | 67 (81)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 30 (36) | 22 (25)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 24 (27) | 13 (18)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 32 (37) | 16 (16)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 13 (13) | 6 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 17 (18) | 27 (28)
MYALGIA (Musculoskeletal and connective tissue disorders) | 49 (57) | 76 (95)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 27 (29) | 30 (36)
DIZZINESS (Nervous system disorders) | 33 (37) | 20 (22)
DYSGEUSIA (Nervous system disorders) | 37 (41) | 35 (44)
HEADACHE (Nervous system disorders) | 70 (85) | 41 (48)
HYPOAESTHESIA (Nervous system disorders) | 10 (10) | 10 (10)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 56 (60) | 34 (37)
PARAESTHESIA (Nervous system disorders) | 35 (44) | 27 (31)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 40 (44) | 21 (23)
ANXIETY (Psychiatric disorders) | 23 (24) | 18 (20)
DEPRESSION (Psychiatric disorders) | 23 (23) | 11 (11)
INSOMNIA (Psychiatric disorders) | 45 (52) | 35 (38)
DYSURIA (Renal and urinary disorders) | 15 (16) | 5 (5)
POLLAKIURIA (Renal and urinary disorders) | 13 (14) | 2 (2)
AMENORRHOEA (Reproductive system and breast disorders) | 9 (10) | 10 (10)
BREAST PAIN (Reproductive system and breast disorders) | 27 (28) | 20 (21)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 22 (22) | 14 (14)
COUGH (Respiratory, thoracic and mediastinal disorders) | 50 (64) | 27 (30)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 29 (33) | 37 (38)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 54 (61) | 41 (45)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 21 (23)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 22 (22)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 127 (127) | 117 (119)
DERMATITIS (Skin and subcutaneous tissue disorders) | 9 (11) | 12 (12)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 15 (18) | 9 (10)
DRY SKIN (Skin and subcutaneous tissue disorders) | 31 (32) | 28 (29)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 19 (20) | 32 (36)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 31 (31) | 4 (4)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 13 (13) | 21 (22)
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 10 (12) | 6 (6)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (10)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 14 (16) | 15 (15)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 19 (20) | 5 (5)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 11 (11) | 23 (26)
PRURITUS (Skin and subcutaneous tissue disorders) | 36 (42) | 44 (49)
RASH (Skin and subcutaneous tissue disorders) | 46 (52) | 40 (47)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 19 (19) | 3 (3)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 11 (11) | 7 (8)
HOT FLUSH (Vascular disorders) | 69 (77) | 48 (55)
HYPERTENSION (Vascular disorders) | 14 (14) | 12 (14)
LYMPHOEDEMA (Vascular disorders) | 14 (15) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.